CLINICAL TRIAL: NCT01387477
Title: Comparison of Two Strategies of Hypoglycemia Correction in ICU
Brief Title: Lactate to Treat Hypoglycemia
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Institut d'Anesthesiologie des Alpes Maritimes (Other)
Responsible Party: Principal Investigator, Professor C ICHAI, Professor Chair of IAAM, Institut d'Anesthesiologie des Alpes Maritimes
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IAAM 2011-01
Record Dates: First submitted 2011-06-30; First posted 2011-07-04 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Hypoglycemia
Keywords: hypoglycemia; lactate; glucose; ICU
MeSH Terms: conditions — Hypoglycemia | interventions — Lactic Acid; Glucose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lactate (Experimental): infusion of 66 mmol of lactate
  Interventions: Drug: Lactate
- glucose (Active Comparator): infusion of 33 mmol of glucose
  Interventions: Drug: Glucose

INTERVENTIONS:
Drug: Lactate — Infusion of 66 mmol of lactate
  Arms: Lactate
Drug: Glucose — Infusion of 33 mmol of glucose
  Arms: glucose

SUMMARY:
Tight glucose control in intensive care has become a major concern, allowing a reduction in morbidity and mortality. However, its use is limited by the percentage of hypoglycemia which can have severe consequences on the brain. The bispectral index (BIS) is derived from the EEG and measures of brain electrical activity noninvasively. It has already been shown that its value changes according to hypoglycemia and its correction. Furthermore, if the hormonal response to hypoglycemia is well known in healthy and diabetic subjects, it is not the case in ICU patient. The usual treatment of hypoglycemia is based on parenteral infusion of glucose. Btu this can lead to a hyperglycemic rebound that can be deleterious. Lactate is a substrate for gluconeogenesis and an energy substrate during critical situations. It has been shown to improve neurological tests during hypoglycaemia and had cerebral protective properties after a severe head injury. The hypothesis of this study is that sodium lactate is superior than the 30% glucose to correct hypoglycemia in the ICU in terms of glycemic variation, brain function and hormonal response.

ELIGIBILITY:
Inclusion Criteria:

* hypoglycemia under 0.6 g/L

Exclusion Criteria:

* hepatic failure
* hyperlactatemia above 5 mmol/L

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-06 (Estimated); Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Area under the curve of the glycemia | 30 minutes

SECONDARY OUTCOMES:
Bispectral index variation | 60 minutes
Maximum change in glycemia | 30 minutes
Changes in growth hormone and cortisol | 180 minutes
Need for glucose infusion for persistent hypoglycemia | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe Orban, MD, Principal Investigator — Nice University Hospital
Locations (1):
- Réanimation médico-chirurgicale, Nice, France